CLINICAL TRIAL: NCT02208024
Title: Phase I Study to Evaluate the Feasibility of Neoadjuvant Stereotactic Body Radiation Therapy for Resectable Adenocarcinoma of the Pancreatic Head and/or Body
Brief Title: Neoadjuvant Stereotactic Body Radiation Therapy for Resectable Adenocarcinoma of the Pancreatic Head and/or Body
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cincinnati (Other)
Responsible Party: Principal Investigator, Jordan Kharofa, Assistant Professor Radiation Oncology, University of Cincinnati
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCCI-GI-002
Record Dates: First submitted 2014-07-31; First posted 2014-08-04 (Estimated); Results first posted 2021-12-29 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-03

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Stereotactic Body Radiation Therapy (Experimental): 5 fractions of 6.6 Gy delivered twice weekly with each fraction separated by greater than 48 hours over 15 days
  Interventions: Radiation: Stereotactic Body Radiation Therapy

INTERVENTIONS:
Radiation: Stereotactic Body Radiation Therapy
  Other Names: SBRT

SUMMARY:
The purpose of this study is to test the safety of focused radiation (Stereotactic Body Radiation Therapy, SBRT) on patients with pancreatic cancer that will be removed surgically.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years.
* Histologically confirmed pancreatic adenocarcinoma of the head and/or body; at least the majority of the histopathologic specimen must be identified as adenocarcinoma.
* Pancreatic tumors must be considered resectable at time of treatment planning. Definition of resectable: no metastases, less than 180 degree involvement of superior mesenteric vein or portal vein, no involvement of hepatic artery, superior mesenteric artery or celiac artery
* No active infection requiring hospitalization
* Adequate labs
* Life expectancy > 3 months.
* Patient is to have received chemotherapy prior to enrollment. This will typically consist of 3-4 cycles of chemotherapy. Patients will have a 2 week break between last chemotherapy administration and start of SBRT.

Exclusion Criteria:

* Presence of metastatic disease.
* Infections requiring systemic antibiotic treatment.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2014-08-27 (Actual); Primary Completion 2017-10-11 (Actual); Study Completion 2019-05-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Mierzwa, MD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Stereotactic Body Radiation Therapy: 5 fractions of 6.6 Gy delivered twice weekly with each fraction separated by greater than 48 hours over 15 days
  Stereotactic Body Radiation Therapy
Period: Overall Study
Arm/Group | Stereotactic Body Radiation Therapy
Started | 18
Completed | 17
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Stereotactic Body Radiation Therapy
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 16
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Acute (Within 3 Months of Treatment) Grade 3 or Greater Gastrointestinal Toxicity
Description: AEs were reviewed for gastrointestinal toxicity. Toxicities of note include grade 3 or greater gastritis, enteritis, fistula, or ulcer and any other grade 3 or greater gastrointestinal toxicity.
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Stereotactic Body Radiation Therapy
Number analyzed (Participants) | 17
Participants | 0

2. Secondary Outcome: Number of Participants With Late (Greater Than 3 Months After Treatment) Grade 2 Gastritis, Enteritis, Fistula, and Ulcer or Any Other Grade 3 or Greater Gastrointestinal Toxicity
Description: AEs were assessed for gastrointestinal toxicity. Toxicities of note include grade 2 or greater gastritis, enteritis, fistula, or ulcer and any other grade 3 or greater gastrointestinal toxicity.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Stereotactic Body Radiation Therapy
Number analyzed (Participants) | 17
Participants | 0

3. Secondary Outcome: Local Progression Free Survival
Description: Local tumor progression will be defined as >=20% increased size on CT scan compared to a CT. scan from prior to treatment. Distant progression will be defined as any new tumor found outside of the pancreas or periampullary region on CT scan. Local and/or distant progression will be evaluated by both PET/CT (if available) and CT scan as deemed by treating physician.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Stereotactic Body Radiation Therapy
Number analyzed (Participants) | 17
Participants | 13

4. Secondary Outcome: Metastasis Free Survival
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Stereotactic Body Radiation Therapy
Number analyzed (Participants) | 17
Participants | 11

5. Secondary Outcome: Overall Survival
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Stereotactic Body Radiation Therapy
Number analyzed (Participants) | 17
Participants | 14

ADVERSE EVENTS:
Time Frame: AEs will be collected up to 12 months after the start of treatment.
Description: The definition does not differ from the definitions used from the clinicaltrial.gov definitions.
Arm/Group | Stereotactic Body Radiation Therapy
All-Cause Mortality (participants affected / at risk) | 11/17
Serious Adverse Events (participants affected / at risk) | 2/17
Other Adverse Events (participants affected / at risk) | 8/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stereotactic Body Radiation Therapy (N=17)
Thromboembolic event (Vascular disorders) | 1 (2)
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stereotactic Body Radiation Therapy (N=17)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Appendicitis perforated (Infections and infestations) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Upper respiratory infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Weight loss (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-04-15): https://cdn.clinicaltrials.gov/large-docs/24/NCT02208024/Prot_SAP_000.pdf